CLINICAL TRIAL: NCT06369506
Title: Classification of Gingival Phenotype at Different Landmarks
Brief Title: Evaluation of Gingival Thickness Measurement at Different Anatomical Landmarks
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Sude Yildirim, Research assistant, Ondokuz Mayıs University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: PYO.DIS.1904 Protocol ID:4467
Record Dates: First submitted 2024-04-09; First posted 2024-04-17 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Gingival Thickness
Keywords: gingiva; gingival phenotype; gingival thickness

STUDY DESIGN:
Intervention Model Description: Participants were divided into two different classifications: "thin" and "thick". The first classification was made by measuring the GT of the point corresponding to the base of the gingival sulcus. GT was defined as thin if ≤1 mm, and thick if >1 mm. In the second classification, GT was measured from three different points. And according to the average GT of three points, they were equally classified as "thin" and "thick".
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gingival Phenotype Classification 1 (Active Comparator): According to the GT of the point corresponding to the GT of the gingival sulcus base
  Interventions: Diagnostic Test: GTmeasurement
- Gingival Phenotype Classification 2 (Active Comparator): According to the average GT of three points
  Interventions: Diagnostic Test: GTmeasurement

INTERVENTIONS:
Diagnostic Test: GTmeasurement — GT was measured from the point corresponding to the base of the gingival sulcus and 1 mm and 2 mm apical to this point. If the GT was ≤1 mm, it was considered a thin phenotype, and if it was >1 mm, it was considered a thick phenotype.

SUMMARY:
In this study, the point at which gingival thickness (GT) should be measured was investigated. Measurements were made from three different points. It was classified as thin and thick in two ways, according to the average of these three different points and the point corresponding to the base of the gingival groove, which is frequently used in the literature. And these two classifications were compared.

DETAILED DESCRIPTION:
The morphology of the soft tissue around the teeth (buccolingual GT and keratinized gingival width) is defined as the "gingival phenotype". One of the most important considerations when assessing gingival phenotype is the objective quantification of GT, and various methods have been used to measure GT. However, there is no clear consensus in the literature regarding the anatomical point where GT is measured in the buccal region. For this reason, it is thought that measurements made from different points also affect the classification of gingival phenotype. The aim of this study was to investigate the cut-off values in clinical parameters according to the average GT value of different measurement points and the GT value at a single point.

The study was designed as cross-sectional study. Participants were divided into two groups based on thin and thick gingival phenotypes in two different classifications. The first classification was based on the GT measurement taken from the base of the gingival sulcus, while the second classification was based on the average of GT measurements taken from three points (base of the gingival sulcus, 1 mm apical to the base of the gingival sulcus, and 2 mm apical to the base of the gingival sulcus. Other clinical and morphological parameters of the participants, who were divided into two groups (thin and thick) according to these classifications, were also measured with a digital caliper and periodontal probe. These parameters are keratinized gingival width (KGW), gingival groove depth (SD), crown width (CW), crown length (CL), crown width/crown length (CW/CL), papilla height (PH), gingival angle (GA). is. Among these parameters, the unit of measurement for GA is angle. CW/CL is the ratio. Other measurements were measured in mm. For all parameters, cut-off values were obtained through statistical measurements made according to two classifications. And these measurements were compared. In addition, the compatibility of the GT measurements of the three points with each other was also examined.

Participants Ondokuz Mayis University's Clinical Research Ethics Board approved the consent form and study protocol (210/2021). Participants with 1195 teeth sites, were enrolled in the study from September 2022 to August 2023. Participants were recruited from University Ondokuz Mayis included patients, dental/ hygiene students. A single calibrated examiner (SY) performed all clinical and morphological measurements.

ELIGIBILITY:
Inclusion Criteria:

* Non-smokers
* Healthy and normal periodontia
* Participants with no evidence of dental caries, crown shape alterations, or restorations affecting the occlusal edge in the teeth
* Presence of at least one tooth representing the anterior, molar and premolar regions in the maxillary and mandibular segments

Exclusion Criteria:

* Presence of gingival recession
* Presence of restorations affecting the crown shape and the occlusal edge of the tooth
* Using any medication that may affect the thickness of periodontal soft tissues (cyclosporine A, phenytoin or calcium channel blockers)
* History of orthodontic treatment
* Craniofacial asymmetry
* History of periodontal surgery
* Presence of abrasion or attrition in the incisal area of the teeth

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-09-10 (Actual); Primary Completion 2023-08-05 (Actual); Study Completion 2023-12-17 (Actual)

PRIMARY OUTCOMES:
Examining the sensitivities and sensitivities of two different gingival phenotype classifications based on three-point average GT measurement and single-point measurement using Receiver Operating Characteristic Analysis (ROC). | 1 month
  Two different classifications compared for determining the gingival phenotype of 50 participants were evaluated for sensitivity and specificity using Receiver Operating Characteristic analysis (ROC). Gingival thicknesses for gingival phenotypes were measured in 1195 teeth. The data were recorded in the SPSS program, and ROC analysis was conducted. The Area Under the Curve (AUC) value is a general measure of classification performance in ROC analysis. AUC value ranges between 0 and 1, with a higher value indicating better performance. The result criterion in ROC analysis is used to evaluate the accuracy and discriminative power of classifications.
Examining the agreement of GT measurements at three different points in 50 patients, 1195 teeth, using Kappa analysis. | 1 month
  50 patients, 1195 teeth in the gingival region were measured in millimeters (mm) using a digital caliper with a precision of 0.001 mm. Kappa analysis was conducted on the collected data. Kappa analysis is used to assess the agreement between two or more measurements or between observers. In this study, the agreement between three points and the average GT value was evaluated using Kappa analysis. Kappa value ranges between -1 and 1: a Kappa value approaching 1 indicates excellent agreement between anatomical points. A negative Kappa value indicates worse agreement than random chance between anatomical points.

CONTACTS AND LOCATIONS:
Overall Officials: Sude Yildirim, DDS, Principal Investigator — Ondokuz Mayis University Department of Periodonthology; Muge Lutfioglu, PHD, Study Director — Ondokuz Mayis University Department of Periodonthology
Locations (1):
- Ondokuz Mayis University Faculty of Dentistry Department of Periodontology, Samsun, Turkey (Türkiye)

REFERENCES:
- [Background] Jepsen S, Caton JG, Albandar JM, Bissada NF, Bouchard P, Cortellini P, Demirel K, de Sanctis M, Ercoli C, Fan J, Geurs NC, Hughes FJ, Jin L, Kantarci A, Lalla E, Madianos PN, Matthews D, McGuire MK, Mills MP, Preshaw PM, Reynolds MA, Sculean A, Susin C, West NX, Yamazaki K. Periodontal manifestations of systemic diseases and developmental and acquired conditions: Consensus report of workgroup 3 of the 2017 World Workshop on the Classification of Periodontal and Peri-Implant Diseases and Conditions. J Periodontol. 2018 Jun;89 Suppl 1:S237-S248. doi: 10.1002/JPER.17-0733. PMID 29926943
- [Derived] Yildirim Bolat S, Lutfioglu M. Evaluation of gingival phenotype: the role of gingival thickness measurements from different vertical gingival levels. Clin Oral Investig. 2025 Jan 25;29(1):87. doi: 10.1007/s00784-024-06143-x. PMID 39856472